CLINICAL TRIAL: NCT00852995
Title: A Phase II Randomized, Double Blind, Placebo Controlled Dose Finding Study Investigating the Efficacy of HP802-247 in Venous Leg Ulcers
Brief Title: Dose Finding Study of HP802-247 in Venous Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 802-247-09-015
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Venous Leg Ulcer; Venous Stasis Ulcers
Keywords: Venous Leg Ulcer (VLU); Venous Stasis Ulcer (VSU); VLU; VSU; Leg Ulcer; Leg Wound
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A - Low Q7D (Experimental): Low dose HP802-247, applied at each visit
  Interventions: Biological: HP802-247
- B - Low Q14D (Experimental): Low dose HP802-247 applied at Visits 1, 3, 5, 7, 9, 11 and Placebo at Visits 2, 4, 6, 8, 10, and 12
  Interventions: Biological: HP802-247
- C - High Q7D (Experimental): High dose HP802-247, applied at each visit
  Interventions: Biological: HP802-247
- D - High Q14D (Experimental): High dose HP802-247, applied at Visits 1, 3, 5, 7, 9, 11 and Placebo at Visits 2, 4, 6, 8, 10, and 12
  Interventions: Biological: HP802-247
- E - Vehicle (Placebo Comparator): Placebo (Vehicle), applied at each visit
  Interventions: Biological: Placebo (Vehicle)

INTERVENTIONS:
Biological: HP802-247 — One dose of HP802-247 consists of 260 microliters (uL) containing keratinocytes and fibroblasts totaling 0.5 x 10-6 power or 5.0 x 10-6 power cells per mL, plus fibrin.
  Arms: A - Low Q7D; B - Low Q14D; C - High Q7D; D - High Q14D
Biological: Placebo (Vehicle) — Placebo (Vehicle) consisting of:
  Component 1 - acellular fibrinogen solution; Component 2 - acellular thrombin solution
  Arms: E - Vehicle

SUMMARY:
This is a 16-week study for subjects with a venous leg ulcer between the knee and ankle. This research is being done to determine the effectiveness of two dosing frequencies and two different concentrations of HP802-247, together with standard care, compared to placebo, plus standard care.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Have a venous leg ulcer (venous etiology)between the knee and ankle, at or above the malleolus.
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Target ulcer duration greater than or equal to 6 weeks but less than or equal to 24 months.

Exclusion Criteria:

* Women who are pregnant or lactating
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies.
* Refusal of or inability to tolerate compression therapy.
* Therapy of the target ulcer with tissue-engineered cell-based skin equivalents within 30 days preceding the Screening Visit.
* Therapy of the target ulcer with topical growth factors within 1 week preceding the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; William Marston, MD, Principal Investigator — University of North Carolina; Robert Kirsner, MD, Principal Investigator — University of Miami; Robert J Snyder, MD, Principal Investigator — Robert J Snyder
Locations (30):
- United States (29):
  - University of AZ College of Medicine, Tucson, Arizona
  - Center for Clinical Research, Castro Valley, California
  - ILD Consulting, Inc., Encinitas, California
  - Vascular Surgery Associates, Los Angeles, California
  - UCSD Wound Treatment and Research Center, San Diego, California
  - University of Miami, Miami, Florida
  - Doctors Research Network, South Miami, Florida
  - Robert J. Snyder, Tamarac, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Passavant Area Hospital, Jacksonville, Illinois
  - Rosalind Franklin University, North Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Johns Hopkins Wound Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New England Sinai Hospital, Stoughton, Massachusetts
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Vincent Giacalone, Emerson, New Jersey
  - St. Luke's Roosevelt Hospital Center, New York, New Jersey
  - Overlook Hospital Wound Healing Program, Summit, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Harrisburg Foot and Ankle Center, Harrisburg, Pennsylvania
  - Center for Advanced Wound Care, Reading, Pennsylvania
  - Arlington Research Center, Arlington, Texas
  - Wound Care Consultants, Dallas, Texas
  - Southwest Regional Wound Care Center, Lubbock, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - Dixie Regional Medical Center's Wound Clinic, St. George, Utah
  - Lake Washington Vascular, LLC, Bellevue, Washington
  - Providence Sacred Heart Medical Center Wound Clinic, Spokane, Washington
- Aging Rehabilitation & Geriatric Care Research Center, London, Ontario, Canada

REFERENCES:
- [Derived] Kirsner RS, Marston WA, Snyder RJ, Lee TD, Cargill DI, Slade HB. Spray-applied cell therapy with human allogeneic fibroblasts and keratinocytes for the treatment of chronic venous leg ulcers: a phase 2, multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2012 Sep 15;380(9846):977-85. doi: 10.1016/S0140-6736(12)60644-8. Epub 2012 Aug 3. PMID 22863328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 34 sites in the US and one in Canada, between June 11, 2009 and May 5, 2011; sites included independent and hospital wound clinics and private practice sites.
Pre-assignment Details: Subjects entered a 2-week run-in; subjects whose wound radius decreased by < 0.349 cm/2weeks and met all other inclusion/exclusion (I/E) criteria were eligible for randomization.
Groups:
- E - HP802-247 Vehicle: Placebo (Vehicle), applied at each visit
  Placebo (Vehicle): Placebo (Vehicle) consisting of:
  Component 1 - acellular fibrinogen solution; Component 2 - acellular thrombin solution
Period: Overall Study
Arm/Group | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D | E - HP802-247 Vehicle
Started | 46 | 43 | 44 | 45 | 50
Completed | 38 | 42 | 39 | 40 | 46
Not Completed | 8 | 1 | 5 | 5 | 4
Not completed — Adverse Event | 1 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 1 | 2
Not completed — Non-Compliance | 0 | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Moved Out of Area | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D | Total
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (14.1) | 61.7 (15.7) | 62.6 (15.4) | 59.8 (15.0) | 61.8 (16.1) | 61.6 (15.2)
Age, Customized [Mean (Full Range); unit: years]
  Female Age | 69.1 [49 to 90] | 61.8 [24 to 87] | 67.7 [33 to 89] | 65.1 [27 to 89] | 69.7 [39 to 94] | 66.5 [24 to 94]
  Male Age | 58.4 [33 to 91] | 61.6 [24 to 88] | 60.1 [28 to 93] | 56.0 [22 to 75] | 58.2 [24 to 80] | 59.0 [22 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 14 | 22 | 20 | 93
  Male | 33 | 26 | 29 | 22 | 25 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 10 | 7 | 13 | 55
  Not Hispanic or Latino | 39 | 32 | 33 | 37 | 32 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 9 | 12 | 8 | 48
  White | 37 | 34 | 30 | 30 | 33 | 164
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 4 | 2 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Average Percent (%) Change From Baseline in the Target Wound Area in Each Treatment Group Over the Twelve-week Double-blind Treatment Period.
Description: For each treatment group the area of each subject's target ulcer was measured on a weekly basis, for up to 12 weeks, or until wound closure, whichever occurred first, using a laser-based wound imaging system in conjunction with software to measure area. An average of the 12 measurements were assessed.
Time Frame: Weekly, over the 12 week treatment period, or until wound closure, which ever occurred first
Population: ITT population.: Subjects who received at least one dose of test article. The primary analysis was performed using a two-way ANCOVA model, which included treatment group (the effect of interest), site, and the baseline target wound area (the covariate), with significance being at P < 0.05.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D | E - HP802-247 Vehicle
Number analyzed (Participants) | 46 | 43 | 44 | 45 | 50
percent change | -77.11 (21.95) | -70.15 (21.66) | -68.14 (26.29) | -72.89 (27.27) | -60.38 (29.79)
Statistical Analysis 1: Comparison: B - Low Q14D vs E - HP802-247 Vehicle; Test type: Superiority or Other; p = 0.00028, t-test, 2 sided
Statistical Analysis 2: Comparison: A - Low Q7D vs E - HP802-247 Vehicle; Test type: Superiority or Other; p = 0.0899, t-test, 2 sided
Statistical Analysis 3: Comparison: D - High Q14D vs E - HP802-247 Vehicle; Test type: Superiority or Other; p = 0.1586, t-test, 2 sided
Statistical Analysis 4: Comparison: C - High Q7D vs E - HP802-247 Vehicle; Test type: Superiority or Other; p = 0.0295, t-test, 2 sided

2. Secondary Outcome: Kaplan-Meier Probability of Non-Closure
Description: This key secondary outcome was the days to wound closure based on a Kaplan-Meier survival analysis.
Time Frame: 14 weeks - the final visit for one subject was delayed by two weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed using the Kaplan-Meier survival procedure, with significance being at P < 0.05.
Measure: Number; unit: Probability of Non-Closure
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
Probability of Non-Closure
  01 week | 1 | 1 | 0.977 | 1 | 1
  02 weeks | 1 | 0.978 | 0.977 | 1 | 0.978
  03 weeks | 0.98 | 0.934 | 0.977 | 0.953 | 0.889
  04 weeks | 0.918 | 0.934 | 0.907 | 0.907 | 0.867
  05 weeks | 0.898 | 0.71 | 0.814 | 0.791 | 0.707
  06 weeks | 0.834 | 0.596 | 0.814 | 0.791 | 0.661
  07 weeks | 0.706 | 0.596 | 0.628 | 0.741 | 0.591
  08 weeks | 0.663 | 0.431 | 0.581 | 0.537 | 0.543
  09 weeks | 0.534 | 0.359 | 0.558 | 0.537 | 0.445
  10 weeks | 0.512 | 0.332 | 0.558 | 0.537 | 0.418
  11 weeks | 0.512 | 0.332 | 0.393 | 0.46 | 0.418
  12 weeks | 0.512 | 0.276 | 0.393 | 0.379 | 0.288
  13 weeks | 0.42 | 0.237 | 0.393 | 0.32 | 0.288
  14 weeks | 0.42 | 0 | 0.393 | 0.32 | 0.288

3. Secondary Outcome: Percent of Change From Baseline in Target Wound Area at Each of the Twelve Double-blind Treatment Weeks.
Description: For each treatment group the area of each subject's target ulcer was measured on a weekly basis, for up to 12 weeks, using a laser-based wound imaging system in conjunction with software to measure area.
Time Frame: Weekly, over the 12 week treatment period, or until wound closure, which ever occurred first
Population: ITT population. Subjects who received at least one dose of test article. The data at each week were analyzed using a two-way ANCOVA model, which included treatment group (the effect of interest), site, and the baseline target wound area (the covariate). Significance was attained at P < 0.05.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
Percent change
  Tx Week 1 | -22.94 (3.97) | -38.88 (4.14) | -27.89 (4.27) | -25.88 (4.26) | -34.97 (4.17)
  Tx Week 2 | -39.94 (4.9) | -58.95 (5.11) | -46.06 (5.26) | -43.69 (5.26) | -49.89 (5.14)
  Tx Week 3 | -47.30 (5.0) | -65.56 (5.22) | -53.5 (5.37) | -55.2 (5.37) | -56.66 (5.25)
  Tx Week 4 | -59.55 (5.28) | -73.46 (5.51) | -62.14 (5.68) | -60.68 (5.68) | -63.92 (5.55)
  Tx Week 5 | -60.54 (5.29) | -79.98 (5.52) | -68.95 (5.68) | -61.87 (5.68) | -72.41 (5.55)
  Tx Week 6 | -63.93 (4.63) | -81.05 (4.83) | -76.01 (4.98) | -74.7 (4.97) | -81.06 (4.86)
  Tx Week 7 | -65.38 (4.64) | -87.22 (4.84) | -79.84 (4.99) | -77.63 (4.98) | -79.81 (4.87)
  Tx Week 8 | -66.62 (5.04) | -83.00 (5.26) | -80.6 (5.42) | -81.58 (5.42) | -81.98 (5.3)
  Tx Week 9 | -69.03 (4.78) | -83.28 (4.99) | -83.96 (5.14) | -84.28 (5.14) | -86.17 (5.02)
  Tx Week 10 | -76.19 (3.39) | -89.65 (3.54) | -85.79 (3.65) | -86.98 (3.65) | -87.74 (3.56)
  Tx Week 11 | -77.05 (3.57) | -89.26 (3.72) | -87.49 (3.84) | -83.37 (3.83) | -87.54 (3.75)
  Tx Week 12 | -80.69 (3.54) | -90.67 (3.69) | -86.87 (3.8) | -84.52 (3.8) | -86.93 (3.72)
Statistical Analysis 1: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .037, ANCOVA — Treatment Week 01
Statistical Analysis 2: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .064, ANCOVA — Treatment Week 02
Statistical Analysis 3: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .161, ANCOVA — Treatment Week 03
Statistical Analysis 4: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .39, ANCOVA — Treatment Week 04
Statistical Analysis 5: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .079, ANCOVA — Treatment Week 05
Statistical Analysis 6: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .069, ANCOVA — Treatment Week 06
Statistical Analysis 7: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .026, ANCOVA — Treatment Week 07
Statistical Analysis 8: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .133, ANCOVA — Treatment Week 08
Statistical Analysis 9: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .089, ANCOVA — Treatment Week 09
Statistical Analysis 10: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .057, ANCOVA — Treatment Week 10
Statistical Analysis 11: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = .127, ANCOVA — Treatment Week 11
Statistical Analysis 12: Comparison: E - HP802-247 Vehicle vs B - Low Q14D vs A - Low Q7D vs D - High Q14D vs C - High Q7D; Test type: Superiority or Other; p = 0.395, ANCOVA — Treatment Week 12

4. Secondary Outcome: Proportion of Subjects Achieving ≥ 50% Decrease in Target Wound Area From Baseline Through Week 13
Description: The area of each subject's target wound was measured at each visit and the proportion of subjects with a decrease in area from baseline ≥ 50% was calculated for each treatment group.
Time Frame: Over the 12 week treatment period or until the wound closed, which ever occurred first.
Population: The non-parametric Cochrane Mantel Haenszel test with adjustment for pooled site was used to examine treatment effects at each time point on the proportion of responders who have an average of ≥50% reduction from baseline in wound area over the treatment period. The test was performed separately for each pair of an active treatment vs. placebo.
Measure: Number; unit: Responders
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
Responders
  Visit 2 | 8 | 17 | 5 | 6 | 13
  Visit 3 | 22 | 29 | 20 | 20 | 21
  Visit 4 | 28 | 34 | 23 | 24 | 31
  Visit 5 | 32 | 38 | 28 | 27 | 34
  Visit 6 | 36 | 40 | 32 | 31 | 36
  Visit 7 | 36 | 39 | 33 | 34 | 42
  Visit 8 | 36 | 43 | 38 | 35 | 41
  Visit 9 | 36 | 43 | 36 | 37 | 41
  Visit 10 | 41 | 40 | 38 | 37 | 40
  Visit 11 | 42 | 44 | 39 | 39 | 43
  Visit 12 | 40 | 42 | 42 | 37 | 41
  Visit 13 | 45 | 45 | 40 | 38 | 40
Statistical Analysis 1: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0133, Cochran-Mantel-Haenszel — Visit 02
Statistical Analysis 2: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.3839, Cochran-Mantel-Haenszel — Visit 02
Statistical Analysis 3: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.5721, Cochran-Mantel-Haenszel — Visit 02
Statistical Analysis 4: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.232, Cochran-Mantel-Haenszel — Visit 02
Statistical Analysis 5: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0787, Cochran-Mantel-Haenszel — Visit 03
Statistical Analysis 6: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.7919, Cochran-Mantel-Haenszel — Visit 03
Statistical Analysis 7: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.6881, Cochran-Mantel-Haenszel — Visit 03
Statistical Analysis 8: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.9832, Cochran-Mantel-Haenszel — Visit 03
Statistical Analysis 9: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0466, Cochran-Mantel-Haenszel — Visit 04
Statistical Analysis 10: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.8435, Cochran-Mantel-Haenszel — Visit 04
Statistical Analysis 11: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.8743, Cochran-Mantel-Haenszel — Visit 04
Statistical Analysis 12: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.2884, Cochran-Mantel-Haenszel — Visit 04
Statistical Analysis 13: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0387, Cochran-Mantel-Haenszel — Visit 05
Statistical Analysis 14: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.8461, Cochran-Mantel-Haenszel — Visit 05
Statistical Analysis 15: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.9574, Cochran-Mantel-Haenszel — Visit 05
Statistical Analysis 16: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.2994, Cochran-Mantel-Haenszel — Visit 05
Statistical Analysis 17: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.1024, Cochran-Mantel-Haenszel — Visit 06
Statistical Analysis 18: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.8759, Cochran-Mantel-Haenszel — Visit 06
Statistical Analysis 19: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.9008, Cochran-Mantel-Haenszel — Visit 06
Statistical Analysis 20: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.4618, Cochran-Mantel-Haenszel
Statistical Analysis 21: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.2439, Cochran-Mantel-Haenszel — Visit 07
Statistical Analysis 22: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.749, Cochran-Mantel-Haenszel — Visit 07
Statistical Analysis 23: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.3749, Cochran-Mantel-Haenszel — Visit 07
Statistical Analysis 24: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel — Visit 07
Statistical Analysis 25: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0078, Cochran-Mantel-Haenszel — Visit 08
Statistical Analysis 26: Comparison: A - Low Q7D; Test type: Superiority or Other; p = 0.07, Cochran-Mantel-Haenszel — Visit 08
Statistical Analysis 27: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.208, Cochran-Mantel-Haenszel — Visit 08
Statistical Analysis 28: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.0413, Cochran-Mantel-Haenszel — Visit 08
Statistical Analysis 29: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0054, Cochran-Mantel-Haenszel — Visit 09
Statistical Analysis 30: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.2031, Cochran-Mantel-Haenszel — Visit 09
Statistical Analysis 31: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.0894, Cochran-Mantel-Haenszel — Visit 09
Statistical Analysis 32: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.0288, Cochran-Mantel-Haenszel — Visit 09
Statistical Analysis 33: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.6964, Cochran-Mantel-Haenszel — Visit 10
Statistical Analysis 34: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.59, Cochran-Mantel-Haenszel — Visit 10
Statistical Analysis 35: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.7146, Cochran-Mantel-Haenszel — Visit 10
Statistical Analysis 36: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.5008, Cochran-Mantel-Haenszel — Visit 10
Statistical Analysis 37: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.1235, Cochran-Mantel-Haenszel — Visit 11
Statistical Analysis 38: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.5488, Cochran-Mantel-Haenszel — Visit 11
Statistical Analysis 39: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.4343, Cochran-Mantel-Haenszel — Visit 11
Statistical Analysis 40: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.1114, Cochran-Mantel-Haenszel — Visit 11
Statistical Analysis 41: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.2119, Cochran-Mantel-Haenszel — Visit 12
Statistical Analysis 42: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.0194, Cochran-Mantel-Haenszel — Visit 12
Statistical Analysis 43: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.506, Cochran-Mantel-Haenszel — Visit 12
Statistical Analysis 44: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.2317, Cochran-Mantel-Haenszel — Visit 12
Statistical Analysis 45: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.1144, Cochran-Mantel-Haenszel — Visit 13
Statistical Analysis 46: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.6786, Cochran-Mantel-Haenszel — Visit 13
Statistical Analysis 47: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.7735, Cochran-Mantel-Haenszel — Visit 13
Statistical Analysis 48: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.758, Cochran-Mantel-Haenszel — Visit 13

5. Secondary Outcome: Percentage of Participants With Complete Wound Closure at Each Visit
Description: Treatment groups were compared for the proportion of wounds closed at each weekly visit. For subjects who dropped from the study, their remaining visit values were imputed using LOCF.
Time Frame: Weekly, over the 12 week treatment period
Population: ITT Populations: Subjects who received at least one dose of test article. Analysis was by the Cochrane Mantel Haenszel (CMH) test
Measure: Number; unit: percentage of participants
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
percentage of participants
  Week 01 | 0 | 4.3 | 2.3 | 0 | 2.2
  Week 02 | 2.0 | 8.7 | 2.3 | 7.0 | 11.1
  Week 03 | 8.0 | 23.9 | 9.3 | 14.0 | 20.0
  Week 04 | 10.0 | 30.4 | 18.6 | 20.9 | 28.9
  Week 05 | 16.0 | 37.0 | 25.6 | 23.3 | 33.3
  Week 06 | 24.0 | 47.8 | 39.5 | 27.9 | 40.0
  Week 07 | 28.0 | 52.2 | 41.9 | 39.5 | 44.4
  Week 08 | 36.0 | 58.7 | 41.9 | 48.8 | 51.1
  Week 09 | 36.0 | 60.9 | 55.8 | 48.8 | 55.6
  Week 10 | 40.0 | 60.9 | 60.5 | 53.5 | 62.2
  Week 11 | 40.0 | 65.2 | 58.1 | 60.5 | 64.4
  Week 12 | 46.0 | 69.6 | 58.1 | 65.1 | 64.4
Statistical Analysis 1: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel — Week 04
Statistical Analysis 2: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = .041, Cochran-Mantel-Haenszel — Week 04
Statistical Analysis 3: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = .017, Cochran-Mantel-Haenszel — Week 05
Statistical Analysis 4: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .011, Cochran-Mantel-Haenszel — Week 06
Statistical Analysis 5: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .014, Cochran-Mantel-Haenszel — Week 07
Statistical Analysis 6: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .029, Cochran-Mantel-Haenszel — Week 08
Statistical Analysis 7: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .021, Cochran-Mantel-Haenszel — Week 09
Statistical Analysis 8: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = .041, Cochran-Mantel-Haenszel — Week 10
Statistical Analysis 9: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .044, Cochran-Mantel-Haenszel — Week 10
Statistical Analysis 10: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .013, Cochran-Mantel-Haenszel — Week 11
Statistical Analysis 11: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = .024, Cochran-Mantel-Haenszel — Week 11
Statistical Analysis 12: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .027, Cochran-Mantel-Haenszel — Week 12

6. Secondary Outcome: Target Ulcer Pain Was Measured Using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects Marked Their Pain Level on a 100 mm Horizontal Line, With a Short Vertical Line Across the Scale, 0 Denoting no Pain and 100mm the Maximum Pain.
Description: Target ulcer pain was measured using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects marked their pain level on a 100 mm horizontal line, with a short vertical line across the scale, 0 denoting no pain and 100mm the maximum pain. Each weekly measurement is reported as the average of all subjects scores at each week per treatment group.
Time Frame: Weekly, over the 12 week treatment period
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed by an ANCOVA, adjusted for site and baseline score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
units on a scale
  Baseline | 30.82 (31.22) | 21.11 (25.23) | 28.6 (21.77) | 29.84 (26.36) | 25.47 (27.7)
  Week 03 | 21.68 (25.01) | 13.37 (18.61) | 16.87 (19.22) | 18.81 (22.15) | 14.42 (18.17)
  Week 06 | 10.72 (18.22) | 10.35 (20.43) | 7.35 (13.36) | 12.25 (17.96) | 11.61 (19.03)
  Week 09 | 9.3 (14.96) | 8.85 (18.53) | 4.53 (9.54) | 11.51 (18.29) | 7.01 (13.63)
  Week 12 | 7.95 (13.34) | 6.83 (11.72) | 3.28 (6.83) | 13.22 (20.71) | 6.61 (13.43)

7. Secondary Outcome: Median Time to Achieve Complete Wound Closure, Based on Based on a Kaplan-Meier Survival Analysis, Over the 12-Week Treatment Period From Baseline.
Description: This key secondary outcome was the days to wound closure based on a Kaplan-Meier survival analysis.
Time Frame: 14 weeks - the final visit for one subject was delayed by two weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days to Closure
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Number analyzed (Participants) | 50 | 46 | 43 | 44 | 45
Days to Closure | 71 [57 to NA] — Unable to assess upper limit. The placebo did not reach 50% closure. | 50 [37 to 66] | 64 [43 to NA] — Unable to assess upper limit. The placebo did not reach 50% closure. | 57 [50 to 85] | 57 [43 to 71]
Statistical Analysis 1: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = 0.0211, ANCOVA — P-value for Kaplan-Meier Days to Closure
Statistical Analysis 2: Comparison: E - HP802-247 Vehicle vs B - Low Q14D; Test type: Superiority or Other; p = .0212, Regression, Cox; Hazard Ratio (HR) = 1.83, 95% CI 2-sided [1.09 to 3.04]
Statistical Analysis 3: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.59, ANCOVA
Statistical Analysis 4: Comparison: E - HP802-247 Vehicle vs A - Low Q7D; Test type: Superiority or Other; p = 0.53, Regression, Cox — This is the P-value for the Cox Hazard Ratio; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [.69 to 2.05]
Statistical Analysis 5: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.26, ANCOVA; Kaplan-Meier Days to Closure
Statistical Analysis 6: Comparison: E - HP802-247 Vehicle vs D - High Q14D; Test type: Superiority or Other; p = 0.19, Regression, Cox — This is the P-value for the Cox Proportional Hazard Ratio; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.84 to 2.44]
Statistical Analysis 7: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.10, ANCOVA — P-value for Kaplan Meier Days to Closure
Statistical Analysis 8: Comparison: E - HP802-247 Vehicle vs C - High Q7D; Test type: Superiority or Other; p = 0.06, Regression, Cox — P-value for Cox Proportional Hazard Ratio; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.97 to 2.77]

ADVERSE EVENTS:
Time Frame: The duration of the 12-week treatment period
Description: All subjects randomized to treatment were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each weekly visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | E - HP802-247 Vehicle | B - Low Q14D | A - Low Q7D | D - High Q14D | C - High Q7D
Serious Adverse Events (participants affected / at risk) | 4/50 | 4/46 | 3/43 | 3/43 | 2/45
Other Adverse Events (participants affected / at risk) | 26/50 | 15/46 | 19/43 | 16/44 | 17/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E - HP802-247 Vehicle (N=50) | B - Low Q14D (N=46) | A - Low Q7D (N=43) | D - High Q14D (N=43) | C - High Q7D (N=45)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E - HP802-247 Vehicle (N=50) | B - Low Q14D (N=46) | A - Low Q7D (N=43) | D - High Q14D (N=44) | C - High Q7D (N=45)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
General disorders and administration site conditions (General disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations (Infections and infestations) | 9 (11) | 4 (4) | 8 (9) | 4 (5) | 8 (9)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 4 (5) | 4 (4) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Psychiatric disorders (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous (Skin and subcutaneous tissue disorders) | 14 (26) | 4 (7) | 6 (8) | 7 (17) | 8 (10)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 8 (16) | 3 (4) | 3 (3) | 4 (5) | 5 (5)
Vascular disorders (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less